CLINICAL TRIAL: NCT06134492
Title: Effect of Acyclovir Therapy on the Outcome of Ventilated Patients With Lower Respiratory Tract Infection and Detection of Herpes Simplex Virus in Bronchoalveolar Lavage
Brief Title: Acyclovir in Ventilated Patients With Pneumonia and HSV-1 in BAL
Acronym: HerpMV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Hagel, Principal Investigator, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKSJ0153; BMBF 01KG2301 (Other Grant/Funding Number: Federal Ministry of Education and Research)
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pneumonia, Viral; Ventilator Associated Pneumonia; Community-acquired Pneumonia; Herpes Simplex; Hospital-acquired Pneumonia
Keywords: Pneumonia; Herpes Simplex; Mechanical Ventilation; Aciclovir
MeSH Terms: conditions — Pneumonia, Viral; Pneumonia, Ventilator-Associated; Community-Acquired Pneumonia; Herpes Simplex; Healthcare-Associated Pneumonia; Pneumonia | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Aciclovir therapy
  Interventions: Drug: Acyclovir
- Comparison group (No Intervention): No study-specific treatment measures

INTERVENTIONS:
Drug: Acyclovir — Dosage: 10mg/kg (current) body weight every 8 hours, dose adjustment to renal function according to technical information.
  Mode of administration: intravenous (i.v.)
  Other Names: Aciclovir
  Arms: Treatment group

SUMMARY:
Almost 90 out of 100 people carry herpes simplex viruses (HSV). Once a person has been infected with the herpes viruses, he or she can't get rid of them for the rest of her/his life. For the most part, the viruses are in a dormant state. Only when the immune system is weakened, for example in the case of a serious illness or stress, are the viruses reactivated. They then mainly cause cold sores, which are harmless for healthy people and usually heal without therapy. However, especially in people with a weakened immune system, HSV can also cause serious infections, such as meningitis. In almost every second mechanically ventilated patient in intensive care who has pneumonia, HSV can be detected in the respiratory tract. This is caused by reactivation of the viruses as a result of the severe underlying disease and stress during intensive care therapy. Whether treatment of the herpes viruses (e.g. with acyclovir) is necessary in this situation and helps the patients to cure has not been clarified, especially as acyclovir can also cause side effects such as a deterioration in kidney function. Currently, the physicians decide to treat the herpes viruses in about half of the patients. Several studies have shown that patients for whom the physician decided to treat the viruses survived more often. However, all of these studies looked at the course of the disease only retrospectively and thus are subject to many biases (including physician selection of who receives treatment, missing data). A definitive conclusion as to whether herpesvirus therapy can be recommended cannot be drawn without doubt from these studies. Therefore, the investigators would like to investigate in a randomized controlled trial, i.e. patients are randomly assigned to the experimental (therapy of herpesviruses) or control group (no therapy of herpesviruses), the effect of therapy with acyclovir on survival in ventilated intensive care patients with lower respiratory tract infection (pneumonia) in whom a large amount of HSV was found in the respiratory tract. The goal of the study is to provide clarity on whether therapy will help patients recover.

DETAILED DESCRIPTION:
Herpes-simplex virus (HSV) can be detected in the bronchoalveolar lavage (BAL) in up to 60% of mechanically ventilated (MV) ICU patients with a lower respiratory tract infection (LRTI), depending on the study population and the severity of disease. However, it remains unclear whether the detection represents a harmless viral shedding as a consequence of reactivation, reflecting the severity of the underlying disease and immunoparalysis, or a true clinical infection requiring antiviral therapy. To date, only retrospective studies have investigated the benefit of an antiviral therapy in HSV-positive ICU patients on mechanical ventilation (MV) with LRTI. In a retrospective study and additional meta-analysis on this topic a antiviral treatment was associated with an improved patient outcome, i.e.; lower all-cause hospital mortality (RR 0.74, 95% CI 0.64-0.85) and lower 30-day all-cause mortality (RR 0.75, 95% CI 0.59-0.94; 3 studies). Aim of this study is to determine prospectively in a multicenter, randomized controlled trial whether acyclovir therapy improves outcome in ventilated ICU patients with a LRTI and HSV detection in BAL. Overall, 616 ICU patients with MV and LRTI and HSV1-PCR-detection in BAL (>= 10E3 copies/ml) will be either randomized to receive acyclovir (10mg/kg body weight tid) for 10 days (or discharge from ICU if this is earlier) or no antiviral therapy (control group). Primary efficacy endpoint will be overall survival within 30 days comparing the acyclovir therapy and the control group. Secondary endpoints include ventilation-free days up to day 30, vasopressor-free days until day 30 and safety.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years
2. need for invasive or non-invasive respiratory support
3. PCR HSV-1 detection in BAL (≥ 10^3 copies/ml)
4. Pneumonia (community or healthcare acquired, incl. ventilator-associated pneumonia)
5. declaration of consent by the patient or legal representative

Exclusion Criteria:

1. History of hypersensitivity to acyclovir or valacyclovir or other components of the investigational product.
2. Pregnancy/Lactation
3. Simultaneous participation in another interventional clinical trial
4. Decision to withhold life-sustaining therapies
5. Use of a virostatic agent (i.v. or p. os) with activity against herpes simplex (acyclovir, valacyclovir, famciclovir/penciclovir, brivudine, cidofovir, foscarnet) for therapeutic or prophylactic reasons at the time of randomization.
6. Solid organ transplantation, stem cell transplantation
7. Neutropenia (absolute neutrophil count <1500/μl (<1.5 × 109 /l)
8. Previous study participation in HerpMV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
mortality (survival status) | day 30
  survival status

SECONDARY OUTCOMES:
Ventilation-free days | day 30
  days without mechanically ventilation via endotracheal tube, incl. tracheostoma
Vasopressor-free days | day 30
  days without continuous vasopressor administration > 1h/day
Delta SOFA score (Sepsis-related Organ Failure Assessment Score) | Baseline - Day 10 or EOT if this event occurs earlier
  Each of six organ systems receive a score ranging from 0 (normal) to 4 (most abnormal), with a minimum SOFA score of 0 and a maximum SOFA score of 24
Delta SOFA sub-score kidney (Sepsis-related Organ Failure Assessment Score) | Baseline - Day 10 or EOT if this event occurs earlier
  Sub-score for kidney function, the score ranges from 0 (normal) to 4 (most abnormal)
Delta GFR value | Baseline - Day 10 or EOT if this event occurs earlier
  GFR value
Length of stay in ICU | day 30
  days LOS in ICU
Length of stay in Hospital | day 30
  days LOS in hospital
Cost of intervention | up to day 90
  ICU and hospitalization days + acyclovir
Days without delirium/coma | Until day 10 or until EOT if this event occurs earlier
  based on CAM-ICU / RASS
Microbiological cure (EOT) | At day 10 or day of EOT if this event occurs earlier
  Percent of participants with HSV eradication (PCR testing negative) in blood and respiratory tract
mortality (survival status) | 90 days
  survival status
mortality (survival status) | 180 days
  survival status
Quality of life (EQ-5D-5L) | Measurement at day 10 or EOT if this event occurs earlier, day 30, day 90, and day 180
  EuroQuality of Life Five Dimensions (EQ-5D-5L), the descriptive system comprises five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT and ANXIETY / DEPRESSION), with five response levels: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems.
Incidence SAEs | From time of randomization until day 10 or EOT if this event occurs earlier
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Locations (25):
- Germany (25):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Klinikum der Ludwig-Maximilian-Universität München, München, Bavaria
  - Klinikum rechts der Isar, München, Bavaria
  - Klinikum Nürnberg, Campus Nord, Nuremberg, Bavaria
  - Klinikum Nürnberg, Campus Süd, Nuremberg, Bavaria
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - RoMed Klinikum Rosenheim, Rosenheim, Bavaria
  - Marien Hospital Herne, Universitätsklinikum der Ruhr-Universität Bochum, Herne, Nordreihn-Westfalen
  - Evangelisches Klinikum Bethel, Bielefeld, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Köln AöR, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck, Schleswig-Holstein
  - Universitätsklinikum Jena, Jena, Thuringia
  - Evangelisches Klinikum Bethel, Bielefeld
  - Universitätsklinikum Hamburg Eppendorf, Hamburg

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a journal indexed in MEDLINE and CTIS; there are no publication restrictions. After publication, deidentified, individual participant data that underlie this trial, along with a data dictionary describing variables in the dataset, will be made available to researchers whose proposed purpose of use is approved by the Trial Management Team.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication

REFERENCES:
- [Derived] Hagel S, Brillinger N, Decker S, Deja M, Ertmer C, Fiedler S, Franken P, Heim M, Weigand MA, Zarbock A, Pletz MW; SepNet Critical Care Trials Group. Effect of acyclovir therapy on the outcome of mechanically ventilated patients with lower respiratory tract infection and detection of herpes simplex virus in bronchoalveolar lavage: protocol for a multicentre, randomised controlled trial (HerpMV). BMJ Open. 2024 Apr 25;14(4):e082512. doi: 10.1136/bmjopen-2023-082512. PMID 38670599
- See also: Study protocol — https://bmjopen.bmj.com/content/14/4/e082512